CLINICAL TRIAL: NCT04246203
Title: Prognostic Role of Circulating Tumor DNA in Resectable Pancreatic Cancer
Acronym: PROJECTION
Status: Active, not recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Benedikt Westphalen, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: ML40429
Record Dates: First submitted 2020-01-26; First posted 2020-01-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: Patients are allocated to group A according to preoperative presence of detectable ctDNA.
  Interventions: Other: Liquid Biopsy
- Group B: Patients are allocated to group B according to preoperative absence of detectable ctDNA.
  Interventions: Other: Liquid Biopsy

INTERVENTIONS:
Other: Liquid Biopsy — 17-20 ml of blood will be collected prior of surgery and within 14 days before start of adjuvant chemotherapy.

SUMMARY:
This is a non-randomized, multicenter, non-interventional study in patients with resectable PDAC. The patients are allocated to two observation groups according preoperative presence of ctDNA (Group A) or absence of detectable ctDNA (Group B) as determined in a liquid biopsy. After successful surgery of their pancreatic tumor and completion of local histological evaluation, tissue samples will be analyzed with regard to their mutational status with. Within 14 days before start of adjuvant tumor therapy another liquid biopsy will be taken to reassess the level of ctDNA after surgery.

Patients will be monitored for disease recurrence according to harmonized, institutional standards using clinical, laboratory and (cross-sectional) imaging modalities. Accordingly, patients will be assessed every three months in the first eighteen months after surgery and every six months thereafter or based on clinical need for 36 months after the date of surgery Follow up will be documented until occurrence of relapse (or death if death occurs earlier than relapse/progression) for a maximum of 36 months after the date of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years of age
2. Pancreatic mass, suspicious of pancreatic cancer, deemed resectable and resection planned.
3. Patient deemed medically fit for adjuvant chemotherapy by the investigator
4. Patient's legal capacity to consent to study participation
5. Signed and dated informed consent to participate in the study

Exclusion Criteria:

1. Non-resectable disease as determined by a local tumor board
2. Metastatic pancreatic disease
3. Previous neoadjuvant chemotherapy
4. Previous neoadjuvant radiotherapy
5. Histology other than PDAC such as acinar, neuroendocrine, mixed histology etc. in the resection specimen
6. Malignant disease other than PDAC within previous year (exception: patients with adequately treated and completely resected basal cell or squamous cell skin cancer; in situ cervical, breast or prostate cancer within previous year may be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic mass, suspicious of pancreatic cancer and deemed resectable will be prospectively enrolled in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
DFS | Follow up will be 36 months after surgery.
  Comparison of disease-free survival (DFS) of patients with preoperative presence of ctDNA (Group A) and absence of ctDNA (Group B)

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Westphalen, Principal Investigator — LMU Munich
Locations (6):
- Germany (6):
  - Ludwig Maximilians University Munich, Munich, Bavaria
  - Charité - Universitätsmedizin Berlin, Berlin
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Technische Universität München, Munich
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Undecided